CLINICAL TRIAL: NCT03981107
Title: A Randomized Trial Comparing Survival After of a Simplified Form of Cardiopulmonary Resuscitation (CPR) Consisting of Compressions Only Compared to CPR With Compressions and Rescue Breaths
Brief Title: Compression Only CPR Versus Standard CPR in Out-Of-Hospital Cardiac Arrest - A Randomized Survival Study
Acronym: TANGO2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Heart Lung Foundation (Other); The Swedish Research Council (Other Government); SOS Alarm (Unknown); Azienda Regionale Emergenza Urgenza - AREU Lombardia (Other)
Responsible Party: Principal Investigator, Jacob Hollenberg, Professor, Head of research - Centre For Resuscitation Science., Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCT3
Record Dates: First submitted 2019-06-05; First posted 2019-06-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Cardiac Arrest; Cardiopulmonary Resuscitation
Keywords: Cardiopulmonary Resuscitation; Chest compressions only CPR; Dispatcher assisted CPR; Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Intervention Model Description: Randomized, 1:1, open label, multicenter trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Because of the inherent logistical problems with blinding of CPR techniques for dispatchers, the trial is considered as an "open labeled" trial. Treatment allocation will, however, be blinded in data management and at follow-up, for personnel treating the patients at the hospitals and for all responsible researchers. Allocation concealment will be preserved.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chest Compression Only CPR (CO-CPR) (Experimental): Instructions from a dispatcher at the dispatch center to trained bystanders to perform CO-CPR with chest compressions only.
  Interventions: Other: Chest Compression Only CPR (CO-CPR) performed by trained bystanders after instructions from dispatchers
- Standard CPR (S-CPR) (Active Comparator): Instructions from a dispatcher at the dispatch center to trained bystanders to perform S-CPR with chest compressions and rescue breaths in a 30:2 ratio.
  Interventions: Other: Standard CPR (S-CPR) performed by trained bystanders after instructions from dispatchers

INTERVENTIONS:
Other: Chest Compression Only CPR (CO-CPR) performed by trained bystanders after instructions from dispatchers — Instructions by dispatcher to bystander to provide CPR with chest-compressions only
  The instructions from the dispatcher in interventional arm include:
  * An ambulance is dispatched and is on it´s way to you
  * Do CPR with chest compressions only
  * Push hard on the chest with a pace of 100/minute without interruptions for rescue breathing.
  Other Names: Chest compression only CPR; Compression only CPR; Hands-only CPR
  Arms: Chest Compression Only CPR (CO-CPR)
Other: Standard CPR (S-CPR) performed by trained bystanders after instructions from dispatchers — Instructions by dispatcher to bystander to provide CPR with chest-compressions and rescue breaths in a ration of 30:2
  The Instructions from the dispatcher in the control arm include:
  * An ambulance is dispatched and is on it´s way to you
  * Do CPR with chest compressions and rescue breathing
  * Push hard on the chest 30 times and give 2 rescue breaths. The pace of the compressions should be 100/minute.
  Other Names: Standard CPR
  Arms: Standard CPR (S-CPR)

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) is one of the leading causes of mortality in the industrialized world. Bystander CPR before arrival of the Emergency Medical Service (EMS) is associated with an increased chance of survival. During the last decade, the best form of bystander CPR has been debated. Chest Compression Only CPR (CO-CPR) has been advocated as a preferable method in situations where the bystander has no previous knowledge in CPR, both because its believed to be equally efficient but also a simplified form of CPR that could lead to a higher incidence of bystander-CPR.

In an initiative to increase CPR rates the American Heart Association has launched public campaigns such as the "hands-only CPR" promoting CO-CPR as an option to S-CPR for adult non-asphyxic cardiac arrest. In the 2015 updates of the European resuscitation council guidelines it states that the confidence in the equivalence between the two methods is not sufficient to change current practice.

Whether CO-CPR leads to a survival rate no worse than, equally effective, or even superior to standard CPR in situations where the bystander has previous CPR training however remains unclear. This clinical question remains unanswered while millions of people are trained in CPR worldwide each year.

The overall purpose with this research project is to investigate whether instructions to perform a simplified form of CPR consisting of compressions only (CO-CPR) to bystanders with prior CPR-training is non-inferior, or better than, standard CPR (S- CPR) in witnessed Out-of-Hospital Cardiac Arrest (OHCA).

DETAILED DESCRIPTION:
This is an interventional, prospective, randomized, 1:1 open label, multicenter trial comparing two different methods of bystander CPR in witnessed cases of OHCA. Since CO-CPR is a simplified form of CPR that could lead to a higher incidence of bystander-CPR by itself a non-inferiority design for the primary outcome has been chosen. Superiority testing will also be performed for the purpose of demonstrating a possible increase in survival with CO-CPR.

Witnessed cases of OHCA with a non-asphyctic aetiology will be the principal study population. According to current guidelines an unresponsive patient with no or agonal breathing is treated as a suspected case of OHCA at the dispatch centre. These cases are eligible for screening for inclusion. If the case is witnessed, the bystander has previous knowledge in CPR and no exclusion criteria are present, the case can be included in the study. If included, it will be randomly assigned to either CO-CPR (intervention) or S-CPR (control).

The intervention consists of instructions from a dispatcher at the dispatch center to bystanders to perform either CO-CPR (intervention) or S-CPR (control).

* Instructions to bystanders on how to perform CO-CPR includes continuous chest compressions without interruptions or rescue breaths.
* Instructions to bystanders on how to perform S-CPR in the control group include information on giving chest compressions and rescue breaths in a 30:2 ratio (like current CPR recommendation state).

This is a national study were all dispatch centers in Sweden participate.

The overall study project is conducted in three different phases:

1. Pre study RUN-IN period, for establishing logistical and technical study procedures (completed)
2. PILOT STUDY, with focus feasibility, logistics and safety (Active, not recruiting)
3. MAIN STUDY will focus on 30 days survival (primary end point) and other important clinical outcomes (secondary outcomes)

Objective pre study RUN-IN period:

In order to test the technical inclusion procedures, logistics, feasibility and data collection a pre-study RUN-IN period started in Stockholm during 2015.

Objective PILOT study:

The aim of the PILOT study is to assess safety and feasibility of the TANGO2 trial design, as well as intermediate clinical outcomes. The TANGO2 trial started recruitment of patients on January 1st 2017 and last patient included on December 31st 2018. All patients from the PILOT study will be included in the MAIN STUDY in a seamless design.

Objective MAIN study:

The aim of the MAIN study is to evaluate whether survival to 30 days following instructions to perform CO-CPR is non-inferior compared to instructions to perform S-CPR bystanders in witnessed OHCA where the bystander has previous CPR training. Secondary and exploratory objectives include the evaluation of neurological favorable survival, return of spontaneous circulation, admission to hospital, long-term survival and other clinical outcome variables as well as evaluations of 30-day survival between CO-CPR and S-CPR in pre-specified subgroups. The MAIN study will include patients from the PILOT phase in a seamless design

Experiences from the pre study RUN-IN period and implications for the PILOT and MAIN studies:

The pre-study RUN-IN period started in Stockholm County in 2015 and analysis were performed during 2016. After continuous technological adjustments, the randomization module was integrated within the computer aided dispatch system and was found to functioned well in the end of 2016. However, during pre-study RUN-IN period, one major obstacle was identified. Due to unexpected technological matters and an unanticipated new organization of the dispatch centers in Sweden only about 15% of the cardiac arrest calls for patients suffering cardiac arrest in Stockholm were actually answered by dispatchers in Stockholm; all other calls were transferred to other dispatch centers throughout Sweden. This meant that the dispatchers had to consider the geographical site of the suspected cardiac arrest and remember if that area was part of the study area. This new organization and logistics, were the call could be made in one area and answered and handled at another site and county during the pre-study RUN-IN period, resulted in a far greatly slower inclusion rate than anticipated and made a correct follow-up of patients unmanageable and unreliable. This made it impossible to conduct a PILOT study in Stockholm only.

As a consequence, a decision was made by the steering committee:

A) To move the start of the PILOT study forward, until completion of the national expansion of the study and not to start inclusion of patients into the PILOT study before January 1st 2017. The new length of the PILOT study was set to two years to assure sufficient inclusion of patients to assess safety in terms of survival to hospital admission.

B) That the PILOT study seamlessly will move on into the MAIN study in an inferentially seamless manner after the PILOT phase inclusion ended on Dec 31 2018. This means that patients from the PILOT study will also be included in the MAIN survival study. The outcomes for the PILOT study were changed to not interfere with the primary endpoint of the main survival study (see below). Inclusion and Exclusion criteria remained unchanged throughout the TANGO2-project.

ELIGIBILITY:
Inclusion Criteria:

* Unconsciousness with no, abnormal or agonal breathing (suspected OHCA)
* The suspected OHCA is witnessed (seen or heard)
* Any Bystander at the scene has previous training in CPR

Exclusion Criteria:

* Age 18 or younger
* Collapse is not witnessed
* Bystander has never been taught CPR. (These bystanders should be instructed to administer CO-CPR in accordance to guidelines)
* Asphyxia, i.e. drowning, strangulation, hanging
* Intoxication or drug overdose
* Pregnancy
* Trauma

Post randomisation exclusion Criteria from data analysis:

* Previous decision that CPR should not be initiated i.e. terminal illness or palliative care
* No Cardiac arrest, other condition (Cases where EMS did not start CPR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3260 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day survival | 1 month
  Survival to 30 days after cardiac arrest

SECONDARY OUTCOMES:
Survival to hospital admission | 1 day
  Survival to admission to hospital
One year survival | 1 year
  Survival to one year after cardiac arrest
Survival with good neurologic outcome at discharge | 30 days
  Survival to hospital discharge with cerebral performance category (CPC) 1-2
Survival with complete neurologically outcome | 30 days
  Survival to hospital discharge with cerebral performance category (CPC) 1

OTHER OUTCOMES:
Proportion of participants found with VT/VF at first rhythm analysis | 1 day
  Proportion of participants found with Ventricular tachycardia (VT) or ventricular fibrillation (VF) at first rhythm analysis by the EMS or by an automated external defibrillator (AED)
Proportion of participants with return of spontaneous Circulation (ROSC) | 1 day
  Proportion of participants with return of spontaneous Circulation
Analysis of primary endpoint (30-day survival) in pre-defined subgroup | 30 days
  Proportion of patients surviving to 30 days after cardiac arrest in subgroups stratified by:
  * Gender
  * Age
  * Cardiac vs non-cardiac cause of OHCA
  * Time to start of CPR
  * Patients with initial shockable rhythm vs initial non-shockable rhythm
  * Call to arrival time of EMS
  * Place of cardiac arrest (at home vs outside home)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Hollenberg, MD, PhD, Principal Investigator — Karolinska Institutet, Department of Medicine Solna; Giuseppe Ristagno, MD, PhD, Study Chair — University of Milan
Locations (2):
- AREU, Agenzia Regionale Emergenza Urgenza, Bergamo, Italy
- SOS Alarm AB, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will be published on group level only

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT03981107/Prot_SAP_001.pdf